CLINICAL TRIAL: NCT02308202
Title: DOXAZOSIN AS A TREATMENT FOR POST TRAUMATIC STRESS SYNDROME
Brief Title: DOXAZOSIN FOR PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Verrico, Associate Professor, Psychiatry Research, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-29283
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: PTSD
Keywords: PTSD; treatment; virtual reality; doxazosin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Doxazosin; Perindopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- doxazosin (Active Comparator): Subjects will be randomized to receive either doxazosin XL or placebo. Participants will receive doses of study medication as over-encapsulated doxazosin XL or placebo dosed once in the morning. Study medication will be initiated as one capsule of doxazosin XL 4 mg or placebo given in the morning. The dose will be titrated up to 16 mg/d doxazosin XL or placebo as follows: Days 1-4: 4mg, Days 5-8: 8mg, Day 9-12: 12 mg, Days 13-16: 16 mg.
  Interventions: Drug: doxazosin
- perindopril (Active Comparator): Subjects will be randomized to receive either perindopril 16mg or placebo for 8 days. Participants will receive doses of study medication as over-encapsulated perindopril or placebo dosed once in the morning.
  Interventions: Drug: Perindopril
- placebo (Placebo Comparator): Subjects will be randomized to receive either doxazosin XL or placebo. Participants will receive placebo for doxazosin XL for 16 days and placebo for perindopril for 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: doxazosin
  Arms: doxazosin
Drug: Perindopril
  Arms: perindopril
Drug: Placebo
  Arms: placebo

SUMMARY:
The aims of this study is to determine the effects of treatment with doxazosin XL 16 mg/d combined with virtual reality (VR) exposure therapy on Post Traumatic Stress Disorder.

The effects of treatment with doxazosin XL 16 mg/d combined with virtual reality (VR) exposure therapy will be assessed in double-blind, placebo-controlled study. The study will enroll 30 participants. The investigators will use a within groups design in which all participants receive both placebo and doxazosin (N=16) with the order counterbalanced across participants. A second group of patients (N=16) will receive both 16mg perindopril and placebo instead of doxazosin/placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Be male OIF/OEF veteran or active duty. Males only are included in this small pilot study because we will not have sufficient sample size to analyze gender effects. Women will be included in subsequent studies
2. Be aged between 18 and 55 years
3. Meet DSM-IV TR criteria for PTSD
4. Meet inclusion criteria for VRE participation
5. Have vital signs as follows: supine blood pressure > 100/65 mm Hg, a seated blood pressure greater than 90/60 mm Hg, and an orthostatic change smaller than20 mm Hg systolic or 10 mm Hg diastolic on standing. Participants should not have hypertension (BP above 150/100)
6. Have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exceptions: (a) total bilirubin must be less than 2x upper limit of normal and ALT, AST, and alkaline phosphatase less than 3× the upper limit of normal and (b) kidney function tests (creatinine and BUN) within normal limits
7. Have a baseline ECG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias
8. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator

Exclusion Criteria:

1. Have any history or evidence suggestive of seizure disorder or brain injury
2. Have neurological or psychiatric disorders, such as psychosis or bipolar illness as assessed by Structural Clinical Interview for DSM disorders (SCID); clinically significant organic brain disease or dementia or Axis I psychiatric illness other than PTSD that would interfere with study; acceptable history of suicide attempts within the past year and/or current suicidal ideation/plan
3. Have evidence of untreated or unstable medical illness including neuroendocrine, autoimmune, renal, hepatic, or active infectious disease
4. Have HIV and are currently symptomatic or are taking antiretroviral medication
5. Have any other illness or condition which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study
6. Dr. Newton (medical supervisor) will review potential participants' prescribed medication to make a final decision on eligibility. We anticipate that participants will be on a wide range of medications prescribed for PTSD. However, these treatments will unlikely interact with the doxazosin effects of this study. We will not ask participants to change their medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are the Subjective Units of Distress Scale (SUDS) and PTSD Checklist (PCL) (m) ratings during VRE Iraq exposure. | 0 and 16 days

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Rodgman C, Verrico CD, Holst M, Thompson-Lake D, Haile CN, De La Garza R 2nd, Raskind MA, Newton TF. Doxazosin XL reduces symptoms of posttraumatic stress disorder in veterans with PTSD: a pilot clinical trial. J Clin Psychiatry. 2016 May;77(5):e561-5. doi: 10.4088/JCP.14m09681. PMID 27249080